CLINICAL TRIAL: NCT00875654
Title: Cell Therapy by Intravenous Injection of Mesenchymal Stem Cells After Stroke
Brief Title: Intravenous Stem Cells After Ischemic Stroke
Acronym: ISIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, AdministrateurCIC, Dr Olivier DETANTE, University Hospital, Grenoble
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCIC 06 25
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Ischemia; Stroke
Keywords: Cell therapy; Stroke; Neuronal Plasticity; Recovery; Mesenchymal Stem Cells; Transplantation
MeSH Terms: conditions — Ischemia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): Control group without intervention nor placebo
- 2 (Experimental): First dose of stem cells
  Interventions: Genetic: Autologous mesenchymal stem cells
- 3 (Experimental): Second dose of stem cells
  Interventions: Genetic: Autologous mesenchymal stem cells

INTERVENTIONS:
Genetic: Autologous mesenchymal stem cells — Intravenous injection of Mesenchymal Stem Cells in a mixing of physiological salt solution/albumin 4% (volume<100ml) less than 6 weeks after stroke
  Arms: 2; 3

SUMMARY:
The main objective of the study is to evaluate feasibility and tolerance of the intravenous injection of autologous mesenchymal stem cells for patients presenting an ischemic stroke (less than 6 weeks).

DETAILED DESCRIPTION:
Stroke is the leading cause of acquired adult disability. Except the hospitalization in stroke units, only thrombolysis has been shown to be efficient to treat acute ischemic stroke in the first three hours after the onset. Increasing brain plasticity after stroke represents an important alternative strategy. Cell therapy provides a functional improvement after cerebral ischemia in rodent models. This "restorative" therapy aims to replace destroyed cerebral tissue with a stem cells graft. Despite these encouraging experiments, we do not know yet the best way of administration of the stem cells, the best dose and the optimal delay of the graft. The pioneer clinical studies failed to reproduce this benefit for patients probably because of the limited number of studied patients. Therefore, more translational studies are needed to improve our knowledge in this promising field. Among different cell sources, mesenchymal (or stromal) stem cells (MSC) derived from bone marrow offer the advantage of arising from a non tumoral and no modified source and are not sources of immunological or ethical problems.

Our research project involves a development of cell therapy in a phase IIa clinical trial of feasibility and safety in patients (randomised, controlled, open, with 3 parallel groups).

ELIGIBILITY:
Inclusion Criteria:

* right or left carotid ischemic stroke in the 14 previous days, confirmed by MRI.
* Persistent neurological deficit (NIHSS >=7).
* Optimal medical treatment(antithrombotics, antihypertensive, statins).
* General state compatible with a program of functional rehabilitation.

Exclusion Criteria:

* Severe extensive stroke implying vital prognosis.
* Severe persistent neurological deficit (NIHSS > 24).
* Medical history of neurological pathology with a deficit as consequence (Rankin < 3 before stroke).
* Serious psychiatric disease.
* Myocardial infarction less than 3 month old.
* Recurring thromboembolic disease or less than 6 month old.
* Patient with organ transplantation.
* Medical history of infection (HIV,HTLV, HBV, HCV).
* Current immunosuppressive/immunomodulating treatment.
* Medical history of cancer.
* Medical history of chemotherapy.
* Known chronic kidney failure(clearance of creatinin < 90 ml/min/1,73m2).
* Known hepatic failure(diminution of prothrombin level (TP) not corrigiable with vitamin K).
* Obesity hinding the bone-marrow sampling in the iliac crest.
* Pathology implying vital prognosis in the 3 month following stroke.
* Refusal to participate.
* Patient unable to give personally his/her consent.
* Pregnant, parturient and feeding women.
* Woman in age to procreate who could not receive an effective method of contraception during the study.
* Participation to another therapeutic clinical trial or in period of exclusion of a therapeutic clinical study.
* Privation of liberty with a decision of justice or administration, legal protection.
* Non affiliation to social security.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-08; Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
feasibility and tolerance of the intravenous injection of autologous mesenchymal stem cells in patients with carotid ischemic stroke | 2 weeks, 1, 2, 4, 6 months and 1, 2 years

SECONDARY OUTCOMES:
Clinical and functional effects of the intravenous injection of autologous mesenchymal stem cells in patients with carotid ischemic stroke | 2 weeks, 1, 2, 4, 6 months and 1, 2 years
Determination of the most effective dose of stem cells | 2 weeks, 1, 2, 4, 6 months and 1, 2 years
To define the best criteria for a future trial (phase III) | 2 weeks, 1, 2, 4, 6 months and 1, 2 years
To define the best target population for a future study | 2 weeks, 1, 2, 4, 6 months and 1, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Detante, MD, Principal Investigator — University Hospital, Grenoble
Locations (3):
- France (3):
  - Neuroradiology/MRI, University Hospital of Grenoble, Grenoble
  - Stroke Unit, University Hospital of Grenoble, Grenoble
  - Tissular and cell therapy unit, UniversityHospitalof Grenoble, Grenoble

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jaillard A, Hommel M, Moisan A, Zeffiro TA, Favre-Wiki IM, Barbieux-Guillot M, Vadot W, Marcel S, Lamalle L, Grand S, Detante O; (for the ISIS-HERMES Study Group). Autologous Mesenchymal Stem Cells Improve Motor Recovery in Subacute Ischemic Stroke: a Randomized Clinical Trial. Transl Stroke Res. 2020 Oct;11(5):910-923. doi: 10.1007/s12975-020-00787-z. Epub 2020 May 27. PMID 32462427
- [Derived] Hannanu FF, Goundous I, Detante O, Naegele B, Jaillard A. Spatiotemporal patterns of sensorimotor fMRI activity influence hand motor recovery in subacute stroke: A longitudinal task-related fMRI study. Cortex. 2020 Aug;129:80-98. doi: 10.1016/j.cortex.2020.03.024. Epub 2020 Apr 17. PMID 32438012